CLINICAL TRIAL: NCT01611233
Title: Clinical Follow-up of ASR Patients Post-Recall
Brief Title: Massachusetts General Hospital Evaluation of DePuy ASR Hip System
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Depuy, Inc. (Industry)
Responsible Party: Principal Investigator, Orhun Muratoglu, Co-Director, Harris Orthopedics Laboratory, Massachusetts General Hospital
Other Study IDs: 2012P000554
Record Dates: First submitted 2012-05-24; First posted 2012-06-04 (Estimated); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Osteoarthritis
Keywords: metal on metal; hip replacement; ASR; DePuy
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DePuy ASR THA: Adults having received a Depuy ASR metal on metal hip system which is subject to a voluntary recall.

SUMMARY:
DePuy Orthopaedics has issued a voluntary recall of the ASR hip replacement system due to a higher than expected revision rate reported in the England/Wales and Australian national joint registries. There are two types of ASR hip implants used for total hip replacement surgery:

* ASR XL Hip System
* ASR Hip Resurfacing System Massachusetts General Hospital (MGH) in Boston, USA is the study sponsor. MGH is conducting this study with the help of funding from DePuy Orthopaedics. MGH will collect and analyze clinical information from 5,000 subjects around the world. The countries include the United States of America, Australia, South Africa, England, Denmark, Finland and Sweden. MGH will collect and analyze blood test results, X-rays, soft tissue imaging and how well the ASR hips are functioning. MGH will analyze the data annually for 6 years.

The purpose of this study is to follow patients who have the ASR hip system for the next 6 years. The findings of this study may help surgeons to make better informed decisions about monitoring and treatment of patients with ASR hip systems.

DETAILED DESCRIPTION:
Description of the Subject Population:

* Adults who have previously undergone a surgery implanting the DePuy ASR XL Acetabular Hip System or ASR Hip Resurfacing System;
* ASR patients who are already being followed-up by their surgeon at least once a year. This routine follow-up care consists of a clinic visit, blood tests, X-rays and possibly an MRI, Ultrasound or CT scan.

ELIGIBILITY:
Inclusion Criteria

1. Any patient with on-label use of the ASR-XL or ASR component system currently implanted.
2. Able to provide informed consent previously approved by institution's Institutional Review board (IRB) or ethics committee (EC).
3. Able to return for follow-up.
4. Able to complete the required patient reported outcome measures.

Exclusion Criteria

1. Any patient with off-label use indications for the ASR-XL or ASR component system.
2. Any patient who received the ASR-XL implant as a result of a hip resurfacing conversion or a revision THA.
3. Subjects with difficulty in comprehending the Informed Consent Form for any reason.
4. The subject refuses to allow their medical records to be inspected by the Sponsor, representatives of the Sponsor, or the medical office staff.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with DePuy ASR or ASR-XL hip implants
Sampling Method: Non-Probability Sample
Enrollment: 1950 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Implant survival rate after hip arthroplasty using DePuy ASR/ASR-XL implants | From the date of primary hip replacement surgery to the end of the study (up to 6 (+/- 0.5) years after enrollment) or to the date of revision surgery, whichever event occurs first.
  To quantify implant failure rates following voluntary recall of the ASR implant

SECONDARY OUTCOMES:
Incidence of adverse local tissue reaction | On the date of revision surgery, not later than the last, 5 year study follow-up visit (<= 6.5 years after enrollment)
  To quantify incidence of adverse local tissue reaction due to metal debris released from the metal-on-metal ASR implant
Cobalt and Chromium ion levels in serum | Within 24 months before enrollment, at each annual follow-up visit; within 6 months before and then within 6 months after revision surgery (last test results <= 7 years after enrollment date)
  To quantify the levels of cobalt and chromium ions in blood serum for patients with the ASR metal-on-metal implant
Plain radiographic, ultrasound and/or MRI evaluation | Within 24 months before enrollment, each annual follow-up visit and within 6 months before revision surgery (last images results <= 6.5 years after enrollment date)
  To measure component positioning and implant stability in patients with the ASR metal-on-metal implant
Patient reported outcome scores: UCLA, Harris Hip, Case Mix Indicator and EQ-5D | At enrollment and each of the 5 annual follow-up visits ((last surveys <= 6.5 years after enrollment date, unless there is revision surgery, then at the last annual follow-up visit)
  To quantify patient reported variables such as pain, activity, and function using validated questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Orhun Muratoglu, PhD, Principal Investigator — Massachusetts General Hospital
Locations (13):
- United States (5):
  - Northshore University HealthSystem, Glenbrook Hospital, Glenview, Illinois
  - Summit Orthopedics, Woodbury, Minnesota
  - Syracuse Orthopedic Specialists, Syracuse, New York
  - Duke University Medical Center, Durham, North Carolina
  - Texas Hip and Knee Center, Fort Worth, Texas
- Sportsmed Sa, Stepney, South Australia, Australia
- Istituti Ospedalieri Bresciani S.p.A., Brescia, Italy
- South Africa (3):
  - Morningside Medi-Clinic, Bryanston
  - Cape Hip and Knee Practice, Cape Town
  - Westville Hospital, Durban
- United Kingdom (3):
  - Royal Berkshire Hospital, Reading, Berkshire
  - Rotherham NHS Foundation Trust, Rotherham Hospital, Rotherham
  - Sheffield Teaching Hospitals Foundation Trust, Sheffield

REFERENCES:
- [Background] Donahue GS, Lindgren V, Galea VP, Madanat R, Muratoglu O, Malchau H. Are Females at Greater Risk for Revision Surgery After Hip Resurfacing Arthroplasty With the Articular Surface Replacement Prosthesis? Clin Orthop Relat Res. 2016 Oct;474(10):2257-65. doi: 10.1007/s11999-016-4860-x. Epub 2016 Apr 27. PMID 27121872
- [Background] Madanat R, Hussey DK, Donahue GS, Potter HG, Wallace R, Bragdon C, Muratoglu O, Malchau H. Early Lessons From a Worldwide, Multicenter, Followup Study of the Recalled Articular Surface Replacement Hip System. Clin Orthop Relat Res. 2016 Jan;474(1):166-74. doi: 10.1007/s11999-015-4456-x. Epub 2015 Aug 27. PMID 26310677
- [Background] Laaksonen I, Galea VP, Connelly JW, Matuszak SJ, Muratoglu OK, Malchau H. Inferior Radiographic and Functional Outcomes With Modular Stem in Metal-on-Metal Total Hip Arthroplasty. J Arthroplasty. 2018 Feb;33(2):464-469. doi: 10.1016/j.arth.2017.08.042. Epub 2017 Sep 6. PMID 28947371
- [Background] Madanat R, Rolfson O, Donahue GS, Hussey DK, Potter HG, Wallace R, Muratoglu OK, Malchau H. Medial Calcar Erosion Is Associated With Synovial Thickness in Patients With ASR XL Total Hip Arthroplasty. J Arthroplasty. 2016 Nov;31(11):2588-2592. doi: 10.1016/j.arth.2016.04.005. Epub 2016 Apr 13. PMID 27178012
- [Background] Galea VP, Laaksonen I, Matuszak SJ, Connelly JW, Muratoglu O, Malchau H. Mid-term changes in blood metal ion levels after Articular Surface Replacement arthroplasty of the hip. Bone Joint J. 2017 Apr;99-B(4 Supple B):33-40. doi: 10.1302/0301-620X.99B4.BJJ-2016-1250.R1. PMID 28363892
- [Background] Donahue GS, Lindgren V, Galea VP, Madanat R, Muratoglu OK, Malchau H. Risk factors for mid-term revision surgery in patients with articular surface replacement total hip arthroplasty. Hip Int. 2018 Jan;28(1):44-49. doi: 10.5301/hipint.5000524. PMID 28574125
- [Background] Hussey DK, Madanat R, Donahue GS, Rolfson O, Bragdon CR, Muratoglu OK, Malchau H. Scoring the Current Risk Stratification Guidelines in Follow-up Evaluation of Patients After Metal-on-Metal Hip Arthroplasty: A Proposal for a Metal-on-Metal Risk Score Supporting Clinical Decision-Making. J Bone Joint Surg Am. 2016 Nov 16;98(22):1905-1912. doi: 10.2106/JBJS.15.00685. PMID 27852907
- [Background] Madanat R, Hussey DK, Donahue GS, Potter HG, Wallace R, Bragdon CR, Muratoglu OK, Malchau H. The Symmetry of Adverse Local Tissue Reactions in Patients with Bilateral Simultaneous and Sequential ASR Hip Replacement. J Arthroplasty. 2015 Oct;30(10):1794-8. doi: 10.1016/j.arth.2015.04.036. Epub 2015 May 30. PMID 26055146
- [Background] Hussey DK, Madanat R, Donahue GS, Rolfson O, Muratoglu OK, Malchau H. Worse health-related quality of life and hip function in female patients with elevated chromium levels. Acta Orthop. 2016 Oct;87(5):485-91. doi: 10.1080/17453674.2016.1213596. Epub 2016 Jul 26. PMID 27459602